CLINICAL TRIAL: NCT04955587
Title: A Longitudinal Study on Longstanding Complicated Fatigue: Myalgic Encephalomyelitis / Chronic Fatigue Syndrome (ME/CFS), Burnout Syndrome and Post-covid Fatigue
Brief Title: A Longitudinal Study on Longstanding Complicated Fatigue
Status: Active, not recruiting | Type: Observational
Sponsor: Stockholm University (Other)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anna Andreasson, Researcher, Stockholm University
Other Study IDs: EPN2018/1438-31
Record Dates: First submitted 2021-06-14; First posted 2021-07-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Chronic Fatigue Syndrome; Burnout; Covid19
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Burnout, Psychological; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Serum Plasma Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with longstanding complicated fatigue: The participants receive no intervention as part of this study.
- Healthy controls: The participants receive no intervention as part of this study.
- Controls with rheumatic disease: The participants receive no intervention as part of this study.

SUMMARY:
The purpose of the study is to investigate if there are common biopsychosocial vulnerability factors for developing and maintaining fatigue, regardless of the diagnosis. The investigators also believe that subgroups differ in terms of these factors. Participating patients with ME/CFS, burnout syndrome and post-covid fatigue complete a web form at inclusion and after 1, 2, 4, 6, 12, 18 and 24 months. There is no upper limit for the number of participants in the web survey. 150 participants are asked to submit blood samples at a local laboratory in connection with the questionnaires for analysis of inflammatory markers and one urine sample for analysis of nutritional markers. Two control groups are included, 150 patients with rheumatoid arthritis and 50 healthy individuals. The longitudinal design makes it possible to investigate how inflammatory markers, nutritional status, symptom burden, health related quality of life co-vary over time and how work ability and sick leave is affected.

DETAILED DESCRIPTION:
Fatigue is associated with impaired health and severely impaired quality of life and function and there is a need to explore similarities and differences regarding biopsychosocial vulnerability and maintenance factors and consequences in terms of work ability and sick leave in chronic fatigue syndrome (ME / CFS), burnout syndrome (BS) and post-covid fatigue to be able to improve individualized interventions for patient with persistent fatigue. The study examines inflammatory markers, nutritional status, symptom burden, neuropsychiatric conditions, work ability, and sick leave in a longitudinal cohort study over 2 years in patients with different diagnoses who all suffer from persistent fatigue. The hypothesis is that there are common biopsychosocial vulnerability factors for developing and maintaining fatigue, regardless of the diagnosis. The investigators also believe that subgroups can be identified that differ in terms of these factors. The longitudinal design makes it possible to investigate how inflammatory markers, nutritional status, symptom burden, health related quality of life co-vary over time and how work ability and sick leave is affected.

In this study participating patients with ME/CFS, BS and post-covid fatigue complete a web form at inclusion and after 1, 2, 4, 6, 12, 18 and 24 months.

Adult patients registered with a diagnosis of chronic complicated fatigue (ME/CFS or post-covid syndrome) in Take Care (medical record system in Stockholm County, Sweden) or with burnout syndrome from Stressmottagningen Stockholm, will be asked to participate in the study.

* Patients with ME/CFS will be recruited at the Department of Behavior Medicine, Karolinska University Hospital Solna or reached by advertising on social media
* Patients with Post-covid-syndrome will be recruited at Karolinska University Hospital or reached by advertising on social media
* Patients with burnout syndrome will be recruited at Stressmottagningen Stockholm

At baseline, a clinical assessment is performed at the clinic and the patient is asked to leave a venous blood sample and complete a questionnaire. The patients are asked for further blood samples and questionnaires at 1, 2, 4, 6, 12, 18, and 24 months after baseline. 150 participants, 50 in each diagnostic group, are asked to submit blood samples for biobanking at a local laboratory in connection to the questionnaire time points for analysis of inflammatory markers. C-reactive protein (CRP) is analysed at the time of blood samples. They are also asked to give one urine sample for analysis of nutritional markers and to submit a 3-day diet diary for evaluation of dietary intake by a registered dietitian. Participants that only fill out the web-based questionnaire will be included. There is no upper limit for the number of participants in the web survey.

A pilot study with 20 participants with ME/CFS started in 2018 to test and revise the design of the present study. These subjects will be counted in the group of 50 participants with ME/CFS diagnosis when available data allow.

In addition to the participants with persistent fatigue, two control groups are included in the study. 150 patients with rheumatoid arthritis (RA) recruited from the Karolinska University Hospital Rheumatology department and 50 healthy controls. The RA controls fill out the illness generic questionnaires on paper and disease information is taken from the national registry for rheumatic disease and CRP and erythrocyte sedimentation rate (ESR) data is taken from the medical record. The healthy controls follow the same procedure as the patients with persistent fatigue but only fill out the form and give blood samples at one time point.

Research questions:

* Are there differences in patient reported fatigue dimensions, symptom burden including post exertional malaise, sleep disorders, health related quality of life, or inflammatory markers, nutritional markers and dietary intake, between patients with ME/CFS, BS and post-covid fatigue, patients with RA and healthy controls?
* Are inflammatory markers and nutritional status associated with the development/recovery of fatigue and symptom burden in ME/CFS, BS and post-covid fatigue?
* Can different subtypes of patients be identified based on latent factor analysis including fatigue dimensions, symptom profile, neuropsychiatric symptoms, inflammatory markers and nutritional status?
* How does inflammatory markers, nutritional status, symptom burden and health related quality of life influence work ability and sick leave in patients with persistent fatigue over time?

The project group consists of a multidisciplinary team from Stockholm and Linköping universities as well as clinically active at clinics in the two regions who often meet patients with persistent fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis set within Stockholm County of ME/CFS, burnout syndrome or post-COVID-19-syndrome according to the Swedish version of the international classification of disease (ICD)-10
* Control group (rheumatic disease): Diagnosis of rheumatoid arthritis
* Control group (healthy): no diagnosis related to inflammatory disease or fatigue

Exclusion Criteria:

* Organic or neuropsychiatric disease that explain the fatigue among cases diagnosed with ME/CFS, burnout syndrome or post-COVID-19-syndrome according to the Swedish ICD-10

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with a diagnosis of ME/CFS, burnout syndrome or post-COVID-19-syndrome. Control groups with rheumatoid arthritis and healthy controls are also included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue (Multidimensional Fatigue Inventory) | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  The Multidimensional Fatigue Inventory (MFI)-20 assesses five dimensions of fatigue. MFI-20 has an even proportion of positively and negatively worded items that are rated on a 5-point Likert scale. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue. The participants completes the MFI at baseline and after 1, 2, 4, 6, 12, 18 and 24 months.
Change in symptom burden | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  Symptom burden is assessed with a checklist and severity rating of the symptoms in the Canada criteria for ME/CFS. The checklist consists of 25 symptoms rated as present/non present. Severity of present symptoms are rated on a 4-point scale. The total score of 0-125 points with a higher score corresponding to a higher symptom burden. The participants completes this form at baseline and after 1, 2, 4, 6, 12, 18 and 24 months.
Change in Generalized sickness behavior (Sickness questionnaire) | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  The sickness questionnaire assesses symptoms of sickness behavior. 10 items are rated on a 4-point Likert scale, total score ranges from 0-30, the higher the scores the more symptoms. The participants completes the the Sickness questionnaire at baseline and after 1, 2, 4, 6, 12, 18 and 24 months.
Change in health related quality of life (World health organization disability assessment scale) | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  The 12-item scale is summarized to a score of 0-100 and a higher score represents a worse quality of life/functioning. The participants completes WHO disability assessment scale (WHODAS) 2.0 at baseline and after 1, 2, 4, 6, 12, 18 and 24 months.
Change in Inflammatory markers | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  Inflammatory markers will be analysed in collaboration with Linköping University at the end of the study. State of the art methods available at study completion will be used. The participants donate blood sample at baseline and after 1, 2, 4, 6, 12, 18 and 24 months. C-reactive protein is analyzed at the time of blood sampling.
Dietary intake | 6 months
  The participants complete 3 day diet diaries at month 6 that are analysed by a registered dietitian.
Nutritional status | 6 months
  The participants take the Organix Basic test by Nordic Laboratories at month six.
Change in self-reported work ability | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  The participants report their sick leave (in %, higher % higher sick leave) and work ability (in percent, higher percent higher work ability) at baseline and after 1, 2, 4, 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Change in insomnia score (insomnia severity index) | baseline and 1, 2, 4, 6, 12, 18 and 24 months
  Insomnia severity index (ISI) is completed at baseline and after 1, 2, 4, 6, 12, 18 and 24 months. ISI consists of 7 items with a total score ranging from 0 to 28 points, where a higher score corresponds to worse symptoms.
Gastrointestinal symptom burden (gastrointestinal symptom rating scale) | 6 and 18 months
  The participant completes the gastrointestinal symptom rating scale (GSRS-IBS) at 6 and 18 months. The GSRS-IBS includes 13 items that measure the severity of IBS symptoms in five clusters (pain, bloating, constipation, diarrhea, and early satiety) during the last seven days. The items are scored between 1 and 7, where 1 corresponds to "no discomfort at all" and 7 to "very severe discomfort" from the symptom. Total score ranges from 13 to 91, with a higher score corresponding to a higher symptom burden.

OTHER OUTCOMES:
Attention deficit hyperactivity disorder (ADHD) | baseline
  Adult ADHD self-report scale (ASRS). ASRS consists of 18 questions in two parts rated on a 5-point scale where a higher score corresponds to a higher symptom burden. Possible range 0-72 points.
Burnout | baseline
  Shirom-Melamed Burnout Questionnaire (SMBQ)-22 consists of 22 items rated on a 7-point rating scale where a higher total score corresponds to a higher symptom level (range 22-145).
Perfectionism | baseline
  Clinical Perfectionism Questionnaire (CPQ) consists of 12 statements rated on a 4-point Likert scale (range total score 4-48), a higher score corresponds to a higher rate of perfectionism
Attention spectrum disorder (ASD) | baseline
  Ritvo Autism and Asperger Diagnostic Scale (RAADS)-14 consists of 14 statements rated on a 4-point scale with a total score ranging from 0-42, with a higher score corresponding to more severe symptoms.
Presence of hypermobility | baseline
  Participants complete the 5 PQ questionnaire for hypermobility at one time point. The questionnaire includes 5 items answered Yes/no, where 2 or more affirmations are indicative of hypermobility.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Andreasson, A Prof, Principal Investigator — Stockholm University
Locations (1):
- Karolinska University Hospital Solna, dep medical psychology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided